CLINICAL TRIAL: NCT07110948
Title: Long-term Follow-up of Infant Frenotomy/Frenectomy Through Early Childhood
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA CTC-24-0121
Record Dates: First submitted 2025-07-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Ankyloglossia
Keywords: observation
MeSH Terms: conditions — Ankyloglossia | interventions — Oral Frenectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Observational after TT release
  Interventions: Procedure: Tongue tie release

INTERVENTIONS:
Procedure: Tongue tie release — surgical release of tongue tie

SUMMARY:
Ankyloglossia (tongue tie) is an anatomically shortened lingual frenum that impairs appropriate tongue mobility. Initial clinical diagnosis of tongue tie usually begins during infancy with abnormal breastfeeding though not all infants with a tongue tie may exhibit difficulties with breastfeeding. Breastfeeding may be impacted during both the latch and suckle phases. Normal latch requires anterior thrust of the tongue past the mandible with the tongue extending out inferior to the mother's nipple and breast. Normal suckle requires tongue elevation including along the entire palate to form sufficient suction force for milk expression from the breast. An tongue tie limiting anterior mobility may inhibit the ability of the tongue to extend anteriorly for appropriate latch, while a tongue tie limiting mid-tongue elevation may impeded the ability of the tongue to elevate to the palate and form sufficient suction force for appropriate suckle. In either situation, symptoms including poor latch, poor suckle, tiredness, extended feeding time, and for the mother nipple pain, tiredness, and frustration are common.

To our knowledge there is no self-correction for ankyloglossia. The frenum does not disappear or become less restrictive on its own over time. Frequency of functional adaptation is now known. Prevalence of ankyloglossia ranges up to 16% depending on population studied, with averages hovering between 8-12%, with males more likely than females to have a tongue tie. While the prevalence of tongue tie has been studied, there is minimal research on the rate of frenectomy for patients with tongue tie. There is also minimal research on the long term effects of infant frenectomy, including on the indications/need for revision surgery for children experiencing difficulties in feeding/transition to solids, speech, malocclusion and/or sleep and breathing concerns. With the increasing popularity of frenectomy, especially in infants, long term research is necessary. However, due to the lack of existing research an initial observational trial to gather preliminary data to allow for more appropriate planning of future research is indicated.

DETAILED DESCRIPTION:
Ankyloglossia (tongue tie) is an anatomically shortened lingual frenum that impairs appropriate tongue mobility. Initial clinical diagnosis of tongue tie usually begins during infancy with abnormal breastfeeding though not all infants with a tongue tie may exhibit difficulties with breastfeeding. Breastfeeding may be impacted during both the latch and suckle phases. Normal latch requires anterior thrust of the tongue past the mandible with the tongue extending out inferior to the mother's nipple and breast. Normal suckle requires tongue elevation including along the entire palate to form sufficient suction force for milk expression from the breast. An tongue tie limiting anterior mobility may inhibit the ability of the tongue to extend anteriorly for appropriate latch, while a tongue tie limiting mid-tongue elevation may impeded the ability of the tongue to elevate to the palate and form sufficient suction force for appropriate suckle. In either situation, symptoms including poor latch, poor suckle, tiredness, extended feeding time, and for the mother nipple pain, tiredness, and frustration are common.

Tongue tie may also affect swallowing after infancy. Tongue ties can limit tongue extension in the transition from feeding to swallowing and result in poor tongue-jaw dissociation resulting in dysphagia. Restrictions to tongue movement can adversely impact the ability for mastication and lateralization of the bolus leading to greater bolus spread. This can result in poor bolus organization and residue in the vestibules, on the cheeks, and/or retained on tooth surfaces. Limitations to tongue movement, and poor tongue-jaw dissociation, can also create difficulties in recognition of residue in these spaces and the removal of residue from these spaces. Tongue tie can also result in limited mid-tongue elevation, affecting the ability to create appropriate pressure and suction power during the oral phase of swallow to propel the bolus into the pharynx. This may result in compensations to bolus formation to allow for swallowing and/or in residue on the soft palate and/or dorsum of the tongue. Residual infantile swallow from tongue tie may also result in a variety of compensations including anterior or posterior tongue thrusting to provide a relative anchored position to achieve enough tongue pressure in bolus transfer from oral to pharyngeal phases. Poor tongue-jaw dissociation resulting from tongue tie may result in poor tongue muscle tone and endurance, resulting in long term muscular compensations including recruitment of lip, cheek, jaw, and neck muscles for swallowing. This may appear as food aversions, texture preferences and challenges in oral to pharyngeal phase swallowing.

Tongue tie can also adversely affect speech, especially in instances where the tongue tie results in poor tongue-jaw dissociation with significant muscular compensations. Tongue tie restricting anterior movement can limit tongue tip elevation leading to speech sound distortions and/or sound substitutions. Limitations to tongue tip elevation to or near the incisive papillae can lead to tongue tip depression with compensatory use of the blade of the tongue for sound production resulting in a wider column of airflow in speech sounds production. In instances of tongue tie with medial restriction and restrictions to mid tongue elevation, the lateral borders of the tongue may fail to elevate during the production of lingual alveolar and palatal sounds. As the center of the tongue will need to elevate in compensation, this can result in lateral distortions. The tongue tie will also result in elevation of the mandible leading to long term overuse of jaw stabilization muscles. This can display as patients reporting generalized mouth and/or jaw muscle fatigue and/or unclear speech progressively worsening with extended use.

The tongue is also a significant muscle in facial development, occlusion, and airway patency. Restrictions to appropriate tongue mobility are associated with dental malocclusion including dental crowding, Class 2 and Class 3 dental malocclusions, loss of maxillary intercanine space, anterior openbite, and increased mandibular incisor spacing, and gingiva recession. Tongue tie has also been associated with maxillary hypoplasia and soft palate elongation. In some cases, tongue tie revision with appropriate orofacial myofunctional therapy has been shown to help improve existing malocclusion without orthodontic intervention

To our knowledge there is no self-correction for ankyloglossia. The frenum does not disappear or become less restrictive on its own over time. Frequency of functional adaptation is now known. Prevalence of ankyloglossia ranges up to 16% depending on population studied, with averages hovering between 8-12%, with males more likely than females to have a tongue tie. While the prevalence of tongue tie has been studied, there is minimal research on the rate of frenectomy for patients with tongue tie. There is also minimal research on the long term effects of infant frenectomy, including on the indications/need for revision surgery for children experiencing difficulties in feeding/transition to solids, speech, malocclusion and/or sleep and breathing concerns. With the increasing popularity of frenectomy, especially in infants, long term research is necessary. However, due to the lack of existing research an initial observational trial to gather preliminary data to allow for more appropriate planning of future research is indicated.

ELIGIBILITY:
Inclusion criteria

* Infants who have undergone lingual frenectomy
* Infants must have been evaluated by a physician/nurse practitioner/lactation consultant prior to lingual frenectomy.
* referral tracking with AHS PRAC-ID
* mother symptomology documented
* frenal attachment classification documented
* Post-surgical wound management documented

Exclusion criteria

* patients unable to be seen at research clinic annually
* parents unable to take photos of patient's lingual frenum

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants who have had tongue tie release completed with appropriate documentation per protocol Infants may be referred for tongue tie release procedure
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Experienced difficulties in function from limitations to tongue range of motion | 6 years
  The primary objective of this study is to explore the rate at which children who had frenectomy in infancy for the purposes of improving breastfeeding experience difficulties in transition to solids feeding, speech, occlusal development, and/or sleep and breathing necessitating referral for further evaluation related to tongue movement restriction.

CONTACTS AND LOCATIONS:
Locations (1):
- Enjoy Dental, Edmonton, Canada

IPD SHARING:
Plan to Share IPD: No